CLINICAL TRIAL: NCT00436709
Title: A Pilot Study of Bevacizumab With Dose Dense Doxorubicin and Cyclophosphamide (AC) Followed by Dose Dense Nanoparticle Albumin Bound Paclitaxel for the Treatment of Early Stage Breast Cancer
Brief Title: Bevacizumab, Doxorubicin, and Cyclophosphamide Followed By Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Bevacizumab in Treating Patients Who Have Undergone Surgery for Early-Stage Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000529855; MSKCC-06019
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2007-06

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; pegfilgrastim; Cyclophosphamide; Doxorubicin; Taxes; Flow Cytometry; Immunoenzyme Techniques; Immunologic Techniques; Chemotherapy, Adjuvant; Radioimmunodetection

INTERVENTIONS:
Biological: bevacizumab
Biological: pegfilgrastim
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Other: flow cytometry
Other: immunoenzyme technique
Other: immunologic technique
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: immunoscintigraphy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This clinical trial is studying the side effects and how well giving bevacizumab together with doxorubicin and cyclophosphamide followed by paclitaxel albumin-stabilized nanoparticle formulation and bevacizumab works in treating patients who have undergone surgery for early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the cardiac safety of adjuvant concurrent bevacizumab and dose-dense doxorubicin hydrochloride and cyclophosphamide followed by dose-dense paclitaxel albumin-stabilized nanoparticle formulation and maintenance therapy comprising bevacizumab alone in patients with early-stage breast cancer.

Secondary

* Determine the noncardiac toxicity of this regimen in these patients.
* Determine the efficacy of this regimen, in terms of time to tumor recurrence and overall survival, in these patients.
* Explore changes in circulating endothelial cells and circulating tumor cells from pre-treatment levels in patients with no evidence of disease.
* Prospectively explore the use of serial troponin I as a predictor of cardiac toxicity in patients treated with this regimen.
* Prospectively explore the relationship between plasma renin activity and hypertension in patients treated with bevacizumab and chemotherapy.

OUTLINE: This is a nonrandomized, pilot, multicenter study.

Patients receive doxorubicin hydrochloride IV, cyclophophamide IV, and bevacizumab IV over 30-90 minutes on day 1 and pegfilgrastim subcutaneously (SC) on day 2. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1 and pegfilgrastim SC on day 2. Treatment with paclitaxel albumin-stabilized nanoparticle formulation and pegfilgrastim repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising bevacizumab IV over 30-90 minutes on day 1. Treatment with maintenance therapy repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study treatment. Samples are analyzed for circulating endothelial cells (by flow cytomery [FC]), circulating epithelial cells (by immunocytochemistry and FC), troponin I concentrations (by enzyme immunoassay or chemiluminescent microparticle immunoassay), and plasma renin activity (by radioimmunoassay).

After completion of study treatment, patients are followed every 4-6 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer meeting the following criteria:

  * Early-stage disease

    * No stage IV disease
  * More than one synchronous primary breast tumor
  * Lymph node positive OR high-risk lymph node negative
* Candidate for treatment with anthracycline- and taxane-based chemotherapy in the adjuvant setting

  * Must begin therapy within 84 days after the final required surgical procedure
* HER2/neu-negative breast cancer, defined as an immunohistochemistry (IHC) score of 0, 1+ or 2+ and fluorescent in situ hybridization (FISH) not amplified
* No CNS disease (e.g., primary brain tumor or brain metastasis)
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Male or female
* Pre- or post-menopausal
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST or ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio ≤ 1.0
* PT and PTT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* LVEF normal by MUGA scan at baseline
* No significant bleeding within the past 6 months
* No uncontrolled underlying bleeding diathesis
* No nonmalignant systemic disease (e.g., cardiovascular, renal, or hepatic) that would preclude study therapy, including any of the following conditions:

  * Blood pressure > 150/100 mm Hg
  * Unstable angina
  * New York Heart Association class II -IV congestive heart failure
  * Myocardial infarction or stroke within the past 12 months
  * Clinically significant peripheral vascular disease
* No seizures not controlled with standard medical therapy
* No history of stroke
* No known allergy or hypersensitivity to study drugs (prior hypersensitivity to paclitaxel allowed)
* No significant traumatic injury within the past 28 days
* No serious nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No active gastroduodenal ulcer
* No uncontrolled intercurrent illness, including psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior therapy for an ipsilateral or contralateral breast cancer primary allowed provided the following criteria are met:

  * No prior anthracycline therapy
  * Prior hormonal therapy for this previous breast cancer is allowed, but must be stopped during study therapy
  * At least 1 year since prior taxane therapy
* More than 28 days since prior and no concurrent major surgery or open biopsy

  * Anticipated reconstructive surgery (e.g., tissue expander exchange) is allowed during the course of the study (bevacizumab will be held during that time as per protocol guidelines)
* More than 7 days since prior minor surgery, including fine-needle aspiration or core biopsy

  * At least 24 hours since prior indwelling catheter placement
* No prior bevacizumab or other KDR inhibitors (e.g., VEGF Trap, semaxanib, SU6668, vandetanib, vatalanib, AEE788, or IMC-1CII)
* No concurrent full-dose anticoagulation therapy
* No concurrent hormonal therapy as chemoprevention
* Concurrent participation in adjuvant hormone therapy or correlative or companion (e.g., bisphosphonate clinic) studies allowed
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Noncardiac toxicity
Time to tumor recurrence
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Maura N. Dickler, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States